CLINICAL TRIAL: NCT04205695
Title: Comparison of Open-tip End-hole and Close-tip Triple-hole Catheters For Continuous Infraclavicular Analgesia
Brief Title: Comparison of Catheters Orifice Configuration For Continuous Infraclavicular Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Burak Eşkin, Assistant Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/398
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Pain, Postoperative; Catheter Blockage; Anesthesia
Keywords: infraclavicular catheter; upper extremity surgery; Postoperative analgesia; continuous nerve block; Catheter tips configurations
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups; Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: The patients will be randomized to the catheter tip configuration as CEMP (closed-ended multiport catheter) group and OESP (open-ended single port catheter) group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEMP (closed-ended multiport catheter) group (Active Comparator): Infraclavicular closed-ended multiport nerve catheter will be included in the patients undergoing upper extremity surgery for postoperative analgesia
  Interventions: Procedure: CEMP (closed-ended multiport catheter) group; Procedure: Patient-controlled analgesia
- OESP (open-ended single port catheter) group (Active Comparator): Infraclavicular open-ended single port nerve catheter will be included in the patients undergoing upper extremity surgery for postoperative analgesia
  Interventions: Procedure: OESP (open-ended single port catheter) group; Procedure: Patient-controlled analgesia

INTERVENTIONS:
Procedure: CEMP (closed-ended multiport catheter) group — The linear probe will be placed parasagittally at the junction between the clavicle and the choroidal process. After medial to lateral scanning, the branches of the brachial plexus will be seen as posterior, lateral and medial truncus around the axillary artery. Contiplex® FX Non-Stimulating Tuohy Set, 17Ga. x 3½ inches. the Non-Stimulating Needle and the closed-tip multiport catheter will be delivered through the needle and placed at the 6 o'clock position relative to the axillary artery and then secured by forming a tunnel under the skin. After negative aspiration, the location of the catheter will be confirmed by injecting 1-2 ml of local anesthetic under ultrasonic guidance.
  Arms: CEMP (closed-ended multiport catheter) group
Procedure: OESP (open-ended single port catheter) group — The linear probe will be placed parasagittally at the junction between the clavicle and the choroidal process. After medial to lateral scanning, the branches of the brachial plexus will be seen as posterior, lateral and medial truncus around the axillary artery. Contiplex® Non-Stimulating Tuohy Set, 17Ga. x 3½ inches. hhe Non-Stimulating Needle and the Non-Stimulating open-ended catheter will be delivered through the needle and placed at the 6 o'clock position relative to the axillary artery and then secured by forming a tunnel under the skin. After negative aspiration, the location of the catheter will be confirmed by injecting 1-2 ml of local anesthetic under ultrasonic guidance.
  Arms: OESP (open-ended single port catheter) group
Procedure: Patient-controlled analgesia — A patient-controlled analgesic device will be attached to the catheter for postoperative analgesia. continuous peripheral nerve patient-controlled analgesia is as follows: 0.125% bupivacaine; hourly infusion: 4 ml / hour, pca dose (bolus): 5 ml / hour, lock-up time: 30 min, 4-hours limit: 30 ml.

SUMMARY:
Infraclavicular nerve catheter for postoperative analgesia will be included in the 70 adult patients undergoing upper extremity surgery included in the study. These patients will be randomized to the catheter tip configuration as CEMP (closed-ended multiport catheter) group and OESP (open-ended single port catheter) group. Patient controlled analgesia device will be attached to the peripheral nerve catheter of these patients. Demographic data of the number of pushing the button, the amount of bolus dose given, the total dose given in the patient controlled anesthesia device, the need for additional analgesia and the amount, pain scores, complications will be recorded for three days postoperatively. Records will be compared statistically.

DETAILED DESCRIPTION:
Ethics committee approval was received on 10 December 2019, numbered 19/398. The study was planned to include 70 adult patients undergoing upper extremity surgery at Gulhane Training and Research Hospital between 10 December 2019 and February 2020. Continue infraclavicular nerve catheter for postoperative analgesia will be included in the patients included in the study. These patients will be randomized to the catheter tip configuration as CEMP(closed-ended multiport catheter) group and OESP(open-ended single port catheter) group. Patient controlled analgesia device will be attached to the peripheral nerve catheter of these patients. Demographic data of the patients who have placed an infraclavicular catheter and used the catheter successfully for three days postoperatively, the number of pushing the button, the amount of bolus dose given and the total dose given in the patient controlled anesthesia device,the amounts of need for additional analgesia and pain scores(Numeric rating Scale), complications will be recorded. Records will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Score I-III
* upper extremity surgery

Exclusion Criteria:

* emergency surgery,
* secondary surgery,
* chronic pain treatment
* pregnancy,
* any contraindication to peripheral nerve blockade,
* pre-existing peripheral nerve neuropathy,
* allergy to local anesthetics (study medications),
* ASA score ≥ 4,
* neurologic or neuromuscular disease,
* psychiatric disease,
* renal failure,
* hepatic failure,
* NSAID contraindication,
* inability to use a patient controlled analgesia (PCA) device,
* infection at the injection site
* withdrawal of consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
numeric rating scale (NRS) | three days postoperatively
  Pain 0 (no pain) to 10 (worst pain imaginable), ranging from a numeric rating scale (NRS)
data from patient-controlled analgesia (PCA) device | three days postoperatively
  The number of PCA button presses
Data from patient-controlled analgesia (PCA) device | three days postoperatively
  Total amount (ml) of local anesthetic (0.125% bupivacaine) delivered to patient recorded by patient controlled analgesia device.
complications related to opioids | three days postoperatively
  Nausea, Vomiting, Itching, Constipation, Difficulty in urination, Difficulty in Concentration,
the requirement for additional analgesia | three days postoperatively
  Additional analgesic dexketoprofen (trometamol) 50 mg / 2 ml will be administered intravenously as rescue analgesia to patients with an NRS score above 3 and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet B EŞKİN, M.D., Study Director — Gulhane Training and Research Hospital; Ayşegül Ceylan, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)